CLINICAL TRIAL: NCT04772716
Title: Postoperative Complication and Associated Factors Among Patients Operated at Hiwot Fana Specialized University Hospital, Ethiopia
Brief Title: Surgical Outcome at HFSUH
Acronym: POC
Status: Completed | Type: Observational
Sponsor: Haramaya Unversity (Other)
Responsible Party: Principal Investigator, Badhaasaa, Dr, Haramaya Unversity
Other Study IDs: HU,CHMS
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Surgical Outcome
Keywords: outcome
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: operation — The intervention was not decided by the investigator but studied following emergency or elective surgeries undergoing in the system

SUMMARY:
the study was conducted on already intervened hospital patients with surgical management and their final outcome was followed from the chart of the patients.

DETAILED DESCRIPTION:
It was a prospective chart review of operated patient at Hiwot fana specialized hospital for different emergency as well elective surgeries. The study subjects signed informed written consent and their data collected anonymously. the follow up protocol was until discharge from hospital the longest date as 30 days.

ELIGIBILITY:
Inclusion Criteria:

* all operated patients at surgical ward

Exclusion Criteria:

* patients operated at other facilities and transferred here. readmission within a month of discharge

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patient admitted surgical ward and underwent surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
post operative complications | 7 days
  the outcome variable is adichotomous on with no complication and has complictions

CONTACTS AND LOCATIONS:
Locations (1):
- HFSUH, Harar, Harari NS, Ethiopia

IPD SHARING:
Plan to Share IPD: No